CLINICAL TRIAL: NCT05117866
Title: A Multicenter, Single Arm, Open-label Trial of Prasugrel Monotherapy After PCI With the SYNERGY® Stent in Patients With Chronic Coronary Syndrome or Non-ST-elevation Acute Coronary Syndromes
Brief Title: Acetyl Salicylic Elimination Trial JAPAN: The ASET JAPAN Pilot Study
Acronym: ASET-JAPAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meditrix Corp (Industry)
Collaborators: Fujita Health University (Other); Boston Scientific Japan K.K. (Industry); National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Yoshinobu Onuma, Professor of interventional Cardiology, National University of Ireland, Galway, Ireland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR20-023
Record Dates: First submitted 2021-09-16; First posted 2021-11-11 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Chronic Coronary Syndrome; Non ST Segment Elevation Acute Coronary Syndrome
Keywords: prasugrel monotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prasugrel Monotherapy (Experimental): The patients will be loaded with standard dual antiplatelet therapy according to local practice (usually aspirin 81 to 330 mg and clopidogrel 300 mg or prasugrel 20 mg or ticagrelor 180 mg, unless patient is on long-term therapy) prior to the PCI procedure. After PCI, if the results are considered to be satisfactory by the operator based on clinical (e.g. clinical status, ECG, etc.), angiographic and/or findings from intracoronary imaging, only then patients will be enrolled in the study and loaded with prasugrel 20 mg if the patients have not loaded prasugrel prior to PCI or have not taken a maintenance dose of prasugrel before the index PCI. Patients continued with prasugrel only (3.75 mg once a day) for three months in CCS patients and for 12 months in NSTE-ACS patients. Aspirin, clopidogrel, and ticagrelor will be discontinued just after the index procedure.
  Interventions: Drug: prasugrel Monotherapy

INTERVENTIONS:
Drug: prasugrel Monotherapy — Prasugrel Monotherapy according to the local dosage (Loading : 20mg, maintenance: 3.75mg/day)
  Other Names: PCI with the SYNERGY® stent

SUMMARY:
The ASET Japan Pilot study is a multicenter, single arm, open-label trial of single antiplatelet therapy with prasugrel for patients undergoing successful and optimal Percutaneous Coronary Intervention (PCI) for Chronic Coronary Syndrome (CCS) and Non-ST elevation Acute coronary syndrome (NSTE-ACS). The enrollment consists of two phases: i) 200 patients presenting with CCS; ii) 200 patients presenting with NSTE-ACS. The patients will be loaded with standard dual antiplatelet therapy according to local practice (usually aspirin 81 to 330 mg and clopidogrel 300 mg or prasugrel 20 mg or ticagrelor 180 mg, unless patient is on long-term therapy) prior to the PCI procedure. After PCI, if the results are considered to be satisfactory by the operator based on clinical (e.g. clinical status, ECG, etc.), angiographic and/or findings from intracoronary imaging, only then patients will be enrolled in the study and loaded with prasugrel 20 mg if the patients have not loaded prasugrel prior to PCI or have not taken a maintenance dose of prasugrel before the index PCI. Patients continued with prasugrel only (3.75 mg once a day) for three months in CCS patients and for 12 months in NSTE-ACS patients. Aspirin, clopidogrel, and ticagrelor will be discontinued just after the index procedure.

i. CCS patients (phase 1): At the 3-months follow-up visit, prasugrel monotherapy will be replaced by aspirin monotherapy or dual-antiplatelet therapy according to local standard of care. Clinical follow-up with office visit will be performed at 3 months and telephone contacts at 1, and 4 months (final follow-up).

ii. NSTE-ACS patients (phase 2): At the 12-months follow-up visit, prasugrel monotherapy will be replaced by aspirin monotherapy for an observational period of 1 month, followed by antiplatelet treatment according to local practice. Clinical follow-up with office visit will be performed at 1 and 12 months and telephone contacts at 3, 6, 9 and 13 months (final follow-up).

All events will be adjudicated by an independent clinical events committee (CEC).

An independent Data Safety and Monitoring Board (DSMB) will monitor the individual and collective safety of the patients in the study during enrolment of CCS patients and up to 3 months follow-up of CCS patients, and during enrollment of NSTE-ACS patients and up to 12 months follow-up of NSTE-ACS patients (timepoint for primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for CCS patients (phase 1) :

1. Successful PCI with optimal acute stent implantation of one or more SYNERGY stent(s).
2. SYNERGY stent implantation was performed to treat:

   1. at least one de novo lesion with ≥50% diameter stenosis determined by visual assessment in at least one native coronary artery with a vessel size between 2.25 mm and 5.0 mm in diameter.
   2. Non-acute coronary disease, with normal cardiac biomarker values prior to the PCI procedure, and evidences of myocardial ischemia by symptoms or non-invasive/invasive testing.
   3. patients with anatomical SYNTAX Score < 23 prior to PCI
3. Patient has provided written informed consent as approved by the Ethical Committee of the respective clinical site.

Inclusion Criteria for NSTE-ACS patients (phase 2) :

1. Patients with diagnosed Non ST-elevation acute coronary syndrome
2. Patients with anatomical SYNTAX Score < 23 prior to PCI
3. Patient provided written informed consent as approved by the Ethical Committee of the respective clinical site

Post PCI criteria for NSTE-ACS patients

1. Patient is free of angina symptoms at the end of PCI procedure.
2. Successful PCI with optimal acute stent implantation of one or more SYNERGY stent(s).
3. SYNERGY stent implantation was performed to treat at least one de novo lesion with ≥50% diameter stenosis determined by visual assessment in at least one native coronary artery with a vessel size between 2.25 mm and 5.0 mm in diameter.

Exclusion Criteria:

Exclusion Criteria for CCS patients (phase 1):

Candidates will be ineligible for enrolment in the study if any of the following conditions apply:

1. ≤ 20 years of age
2. Unable to give Informed Consent
3. Females of child-bearing potential unless negative pregnancy test at screening and willing to use effective contraception for the duration of treatment with study medication
4. Female who is breastfeeding at time of enrolment
5. Patients concomitantly received any other non-study stent at the same procedure
6. Patients with planned PCI or surgical intervention to treat any cardiac or non-cardiac condition;
7. Previous PCI with any non-SYNERGY stents in the last 6 months
8. Current (same hospitalization) or previous (within 12 months) acute coronary syndrome
9. Patient with following lesion characteristics prior to PCI; Saphenous or arterial graft, in-stent (re)stenosis
10. History of definite stent thrombosis
11. Concomitant cardiac valve disease requiring invasive therapy
12. Atrial fibrillation or other indication for oral anticoagulant therapy
13. Known allergy to aspirin, prasugrel or diagnosed lactose intolerance
14. Acute heart failure
15. Active myocarditis
16. Cardiomyopathy
17. Patient in hemodialysis
18. Treatment in the last 10 days or requirement for ongoing treatment with a strong CYP3A4 inhibitor or inducer;
19. History of stroke or transient ischemic cerebrovascular accident
20. History of intracranial hemorrhage or other intracranial pathology associated with increased bleeding risk
21. Hemoglobin <10 g/dL or other evidence of active bleeding
22. Peptic ulceration documented by endoscopy within the last 3 months unless healing proven by repeat endoscopy
23. Any other condition deemed by the investigator to place the patient at excessive risk of bleeding with prasugrel
24. Participation in another trial with an investigational drug or device
25. Co-morbidity associated with life expectancy <1 year
26. Assessment that the subject is not likely to comply with the study procedures or have complete follow-up
27. Known drug or alcohol dependence within the past 12 months as judged by the investigator

Exclusion Criteria for NSTE-ACS patients (Phase 2):

Candidates will be ineligible for enrolment if any of the following conditions apply:

1. ≤ 20 years of age
2. Unable to give Informed Consent
3. Females of child-bearing potential unless negative pregnancy test at screening and willing to use effective contraception for the duration of treatment with study medication
4. Female who is breastfeeding at time of enrolment
5. Patients concomitantly received any other non-study stent at the same procedure
6. Patients with planned PCI or surgical intervention to treat any cardiac or non-cardiac condition;
7. Previous PCI with any non-SYNERGY stents in the last 6 months
8. Patient with following lesion characteristics prior to PCI; Saphenous or arterial graft, in-stent (re)stenosis
9. History of definite stent thrombosis
10. Concomitant cardiac valve disease requiring invasive therapy
11. Known allergy to aspirin, prasugrel or diagnosed lactose intolerance
12. Atrial fibrillation or other indication for oral anticoagulant therapy;
13. History of stroke or transient ischemic cerebrovascular accident
14. History of intracranial haemorrhage or other intracranial pathology associated with increased bleeding risk
15. Acute heart failure
16. Active myocarditis
17. Cardiomyopathy
18. Patient in hemodialysis
19. Haemoglobin <10 g/dL or other evidence of active bleeding
20. Hemodynamic instability or cardiogenic shock
21. Recurrent or ongoing chest pain refractory to medical treatment
22. Life-threatening arrhythmias or cardiac arrest;
23. Mechanical complications of myocardial infarction
24. Recurrent dynamic ST-T wave changes, particularly with intermittent ST-elevation
25. Peptic ulceration documented by endoscopy within the last 3 months unless healing proven by repeat endoscopy
26. Any other condition deemed by the investigator to place the patient at excessive risk of bleeding with prasugrel
27. Participation in another trial with an investigational drug or device
28. Co-morbidity associated with life expectancy < 1 year
29. Assessment that the subject is not likely to comply with the study procedures or have complete follow-up;
30. Known drug or alcohol dependence within the past 12 months as judged by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Primary Ischemic Endpoint events (CCS) | 3 months
  Composite of cardiac death, target-vessel myocardial infarction (spontaneous >48 hours) or definite stent thrombosis.
Rate of Primary Ischemic Endpoint events (NSTE-ACS) | 12 months
  Composite of cardiac death, target-vessel myocardial infarction (spontaneous >48 hours) or definite stent thrombosis.
Rate of Primary Bleeding Endpoint event (CCS) | 3 months
  BARC 3 or 5 bleeding
Rate of Primary Bleeding Endpoint event (NSTE-ACS) | 12 months
  BARC 3 or 5 bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, MD, PhD, Study Chair — National University of Ireland, Galway; Yoshinobu Onuma, MD, PhD, Study Chair — National University of Ireland, Galway; Takashi Muramatsu, MD, PhD, Principal Investigator — Fujita Health University; Kengo Tanabe, MD, PhD, Principal Investigator — Mitsui Memorial Hospital; Yukio Ozaki, MD, PhD, Principal Investigator — Fujita Health University Hospital and Okazaki Medical Center
Locations (13):
- CORRIB Research Centre for Advanced Imaging and Core laboratoryNational University of Ireland, Galway, Galway, Ireland
- Japan (12):
  - Fujita Health University, Okazaki Medical Centre, Okazaki, Aichi-ken
  - Fujita Health University, Toyoake, Aichi-ken
  - Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Iwate Medical University Hopsital, Morioka, Iwate
  - St. Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - JCHO Hoshigaoka Medical center, Hirakata, Osaka
  - Kinki University Hospital, Faculty of Medicine, Ōsaka-sayama, Osaka
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Mitusi Memorial Hospital, Tokyo
  - St. Luke's international hospital, Tokyo
  - Teikyo University Hospital, Tokyo
  - Toho University Ohashi Medical Center, Tokyo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Masuda S, Muramatsu T, Ishibashi Y, Kozuma K, Tanabe K, Nakatani S, Kogame N, Nakamura M, Asano T, Okamura T, Miyazaki Y, Tateishi H, Ozaki Y, Nakazawa G, Morino Y, Katagiri Y, Garg S, Hara H, Ono M, Kawashima H, Lemos PA, Serruys PW, Onuma Y. Reduced-dose prasugrel monotherapy without aspirin after PCI with the SYNERGY stent in East Asian patients presenting with chronic coronary syndromes or non-ST-elevation acute coronary syndromes: rationale and design of the ASET Japan pilot study. AsiaIntervention. 2023 Mar 15;9(1):39-48. doi: 10.4244/AIJ-D-22-00033. eCollection 2023 Mar. PMID 36936091
- [Result] Muramatsu T, Masuda S, Kotoku N, Kozuma K, Kawashima H, Ishibashi Y, Nakazawa G, Takahashi K, Okamura T, Miyazaki Y, Tateishi H, Nakamura M, Kogame N, Asano T, Nakatani S, Morino Y, Katagiri Y, Ninomiya K, Kageyama S, Takahashi H, Garg S, Tu S, Tanabe K, Ozaki Y, Serruys PW, Onuma Y. Prasugrel Monotherapy After Percutaneous Coronary Intervention With Biodegradable-Polymer Platinum-Chromium Everolimus Eluting Stent for Japanese Patients With Chronic Coronary Syndrome (ASET-JAPAN). Circ J. 2023 May 25;87(6):857-865. doi: 10.1253/circj.CJ-23-0051. Epub 2023 Mar 11. PMID 36908118
- [Result] Masuda S, Tanabe K, Guimaraes PO, Muramatsu T, Ozaki Y, De Martino F, Kozuma K, Garg S, Kotoku N, Ninomiya K, Kageyama S, Lemos PA, Onuma Y, Serruys PW. Prasugrel Monotherapy After Percutaneous Coronary Intervention for Chronic Coronary Syndrome: Insights From ASET Pilot Studies. JACC Asia. 2023 Dec 12;4(3):171-182. doi: 10.1016/j.jacasi.2023.10.007. eCollection 2024 Mar. PMID 38463674
- [Result] Kotoku N, Ninomiya K, Masuda S, Tsai TY, Revaiah PC, Garg S, Kageyama S, Tu S, Kozuma K, Kawashima H, Ishibashi Y, Nakazawa G, Takahashi K, Okamura T, Miyazaki Y, Tateishi H, Nakamura M, Kogame N, Asano T, Nakatani S, Morino Y, Ishida M, Katagiri Y, De Martino F, Tinoco J, Guimaraes PO, Tanabe K, Ozaki Y, Muramatsu T, Lemos PA, Onuma Y, Serruys PW; ASET Japan and ASET Brazil Investigators. Geographic disparity of pathophysiological coronary artery disease characteristics: Insights from ASET trials. Int J Cardiol. 2024 Apr 1;400:131805. doi: 10.1016/j.ijcard.2024.131805. Epub 2024 Jan 23. PMID 38272132
- [Result] Kotoku N, Ninomiya K, Masuda S, O'Leary N, Garg S, Naito M, Miyashita K, Tobe A, Kageyama S, Tsai TY, Revaiah PC, Tu S, Kozuma K, Kawashima H, Ishibashi Y, Nakazawa G, Takahashi K, Okamura T, Miyazaki Y, Tateishi H, Nakamura M, Kogame N, Asano T, Nakatani S, Morino Y, Ishida M, Katagiri Y, Ono M, Hara H, Sotomi Y, Tanabe K, Ozaki Y, Muramatsu T, Dijkstra J, Onuma Y, Serruys PW. Preprocedural physiological assessment of coronary disease patterns to predict haemodynamic outcomes post-PCI. EuroIntervention. 2023 Dec 18;19(11):e891-e902. doi: 10.4244/EIJ-D-23-00516. PMID 37960875
- [Derived] Revaiah PC, Miyashita K, Tsai TY, Bajaj R, Kotoku N, Tobe A, Muramatsu T, Tanabe K, Kozuma K, Ozaki Y, Garg S, Tu S, Dijkstra J, Bourantas CV, Onuma Y, Serruys PW. Segmental post-percutaneous coronary intervention physiological gradients using ultrasonic or optical flow ratio: insights from ASET JAPAN study. Eur Heart J Imaging Methods Pract. 2025 Jan 30;3(1):qyaf017. doi: 10.1093/ehjimp/qyaf017. eCollection 2025 Jan. PMID 39974274
- [Derived] He X, Tsung-Ying T, Revaiah PC, Wykrzykowska JJ, Rosseel L, Sharif F, Muramatsu T, Reiber JH, Garg S, Miyashita K, Tobe A, Tao L, Onuma Y, Serruys PW. Nomogram based on virtual hyperemic pullback pressure gradients for predicting the suboptimal post-PCI QFR outcome after stent implantation. Int J Cardiovasc Imaging. 2024 Dec;40(12):2469-2479. doi: 10.1007/s10554-024-03253-1. Epub 2024 Oct 12. PMID 39395074